CLINICAL TRIAL: NCT04577547
Title: Efficacy of the Dietary Guidelines for Americans and the Physical Activity Guidelines for Americans for Weight Control
Brief Title: Food, Activity and Behavior Study
Acronym: FAB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never started
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: GFHNRC512
Record Dates: First submitted 2020-06-18; First posted 2020-10-08 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Dietary Guidelines (DGA) diet with weight loss (WL) & exercise (Experimental): Menu to provide DGA-recommended food group amounts at a calorie level to promote weight loss with Physical Activity Guidelines for Americans (PAGA)-recommended exercise
  Interventions: Other: DGA diet WL & exercise
- DGA diet with WL & no exercise (Experimental): Menu to provide DGA-recommended food group amounts at a calorie level to promote weight loss with no exercise
  Interventions: Other: DGA diet WL & no exercise
- DGA diet weight maintenance (WM) & exercise (Experimental): Menu to provide DGA-recommended food group amounts at a calorie level to promote weight maintenance with PAGA-recommended exercise
  Interventions: Other: DGA diet WM & exercise
- DGA diet WM & no exercise (Experimental): Menu to provide DGA-recommended food group amounts at a calorie level to promote weight maintenance with no exercise
  Interventions: Other: DGA diet WM & no exercise
- Western diet with WL & exercise (Experimental): Western-type menu to provide a calorie level to promote weight loss with PAGA-recommended exercise
  Interventions: Other: Western diet WL & exercise
- Western diet with WL & no exercise (Experimental): Western-type menu to provide a calorie level to promote weight loss with no exercise
  Interventions: Other: Western diet WL & no exercise
- Western diet WM exercise (Experimental): Western-type menu to provide a calorie level to promote weight maintenance with PAGA-recommended exercise
  Interventions: Other: Western diet WM & exercise
- Western diet WM no exercise (Experimental): Western-type menu to provide a calorie level to promote weight maintenance with no exercise
  Interventions: Other: Western diet WM & no exercise

INTERVENTIONS:
Other: DGA diet WL & exercise — Intake of DGA weight loss 8 day rotating menu & PAGA-recommended exercise
  Arms: Dietary Guidelines (DGA) diet with weight loss (WL) & exercise
Other: DGA diet WL & no exercise — Intake of DGA weight loss 8 day rotating menu & no exercise
  Arms: DGA diet with WL & no exercise
Other: DGA diet WM & exercise — Intake of DGA weight maintenance 8 day rotating menu & PAGA-recommended exercise
  Arms: DGA diet weight maintenance (WM) & exercise
Other: DGA diet WM & no exercise — Intake of DGA weight maintenance 8 day rotating menu & no exercise
  Arms: DGA diet WM & no exercise
Other: Western diet WL & exercise — Intake of Western-type weight loss 8 day rotating menu & PAGA-recommended exercise
  Arms: Western diet with WL & exercise
Other: Western diet WL & no exercise — Intake of Western-type weight loss 8 day rotating menu & no exercise
  Arms: Western diet with WL & no exercise
Other: Western diet WM & exercise — Intake of Western-type weight maintenance 8 day rotating menu & PAGA-recommended exercise
  Arms: Western diet WM exercise
Other: Western diet WM & no exercise — Intake of Western-type weight maintenance 8 day rotating menu & no exercise
  Arms: Western diet WM no exercise

SUMMARY:
The purpose of this research is to test the effects of the Dietary and Physical Activity Guidelines for Americans on health and on eating and exercise behaviors.

DETAILED DESCRIPTION:
The Dietary Guidelines for Americans (DGA), which include the Physical Activity Guidelines for Americans (PAGA), is the primary United States (U.S) government resource for weight control. The researchers propose that chronic, low grade inflammation (CLGI) limits weight control by acting upon physiological and behavioral factors that moderate weight control. Diet and exercise reduce CLGI and provide weight control, but no one has investigated the efficacy of the DGA and PAGA to reduce CLGI, whether reduced CLGI promotes greater weight control, and the moderating roles of physiological and behavioral factors on the association of reduced CLGI with weight control. To accomplish this, the researchers will conduct a 6-month trial in 224 obese adults; a 3-month controlled feeding trial with four dietary arms; 1) DGA with weight loss, 2) Western diet with weight loss,3) DGA diet weight maintenance, 4) Western diet weight maintenance. Each dietary arm will have PAGA-recommended exercise and non-exercise arms. Post-trial is a 3-month weight maintenance period. The primary outcome is change in C-reactive protein (CRP), a marker of CLGI. The results will inform the DGA and PAGA; thereby helping clinicians, public health workers, and policymakers to improve the health of Americans.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI 30.0 kg/m2 - 350 lbs [maximum weight for dual energy x-ray absorptiometry (DXA) machine])
* No contraindications to participate in exercise
* hs-CRP level ≥3.0 and ≤10.0 mg/L or two consecutive measures of >10.0 mg/L measured two weeks apart
* Access to high-speed internet

Exclusion Criteria:

* Taking chronic anti-inflammatory medications
* Being pregnant, lactating, or planning to become pregnant
* Diagnosed eating disorder
* Taking weight loss medication
* Smoking
* Overt hypothyroidism
* Cancer
* Physical conditions that prevent safe exercise
* Liking of <3 out of 10 for all available physical activity modes
* Currently exercising for more than 30 minutes per day >3 days per week
* Unwilling to continue with current exercise routine
* Not willing to comply with all study requirements
* Blood pressure greater than 140/90

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in C-reactive protein (CRP) | Weeks 0, 2, 4, 6, 8, 10, 12, 24
  The effect of diet and exercise on CRP
Relative reinforcing value (RRV) of energy-dense snack foods | Weeks 0,12, 24
  The effect of consuming a healthy DGA style or a Western style diet during weight loss and weight maintenance on the RRV of energy-dense snack food using a computer choice paradigm. For the computer choice paradigm subjects click the mouse button to play a simulated slot machine games to earn points toward receiving a portion of food or being able to do a non-food related sedentary activity (e.g., watching TV).
Relative reinforcing value (RRV) of exercise | Weeks 0,12, 24
  The effect of achieving the DGA recommended amounts of exercise during weight loss and weight maintenance on relative reinforcing value of exercise compared to a sedentary activity alternative using a computer choice paradigm. For the computer choice paradigm subjects click the mouse button to play a simulated slot machine games to earn points toward being able to do a chosen physical activity, such as walking on a treadmill, or a sedentary activity (e.g., watching TV).
Fat and carbohydrate oxidation | Weeks 0,12
  The effect of diet and exercise on carbohydrate and fat oxidation in response to meals and exercise as measured by whole-room calorimetry

SECONDARY OUTCOMES:
Food Cognitive Interference | Weeks 0, 12, 24
  The effect of diet and exercise on food cognitive interference, one of the three cognitive domains of executive function, using a computerized Food Stroop test.
Cognitive flexibility | Weeks 0, 12, 24
  The effect of diet and exercise on cognitive flexibility, one of the three cognitive domains of executive function, using a computerized Trail-Making test B/A.
Working memory | Weeks 0, 12, 24
  The effect of diet and exercise on cognitive flexibility, one of the three cognitive domains of executive function, using the Wisconsin Card Sorting Task.
Inflammation | Weeks 0, 2, 4, 6, 8, 10, 12, 24
  The effect of diet and exercise on plasma pro-inflammatory cytokines (e.g., Il-6, MCP-1, TNF-alpha) and anti-inflammatory cytokines (e.g., IL-10, Soluble TNF receptor I and II)
Change in adipokines | Weeks 0, 2, 4, 6, 8, 10, 12, 24
  The effect of diet and exercise on plasma adipokines (e.g., adiponectin, resistin)
Change in myokines | Weeks 0, 2, 4, 6, 8, 10, 12, 24
  The effect of diet and exercise on plasma myokines (e.g., BDNF, Myostatin, FGF-21, Irisin)
Change in bile acids | Weeks 0, 2, 4, 6, 8, 10, 12, 24
  The effect of diet and exercise on plasma bile acids (i.e., glycocholic acid, glyco-CDCA, glyco-HDCA, hyocholic acid, hyodeoxycholic acid)
Change in blood lipids | Weeks 0, 2, 4, 6, 8, 10, 12, 24
  The effect of diet and exercise on cholesterol, HDL, triglycerides
Change in weight control moderators | Weeks 0,12, 24
  Questionnaires (i.e., three-factor eating questionnaire, reward base eating, food attitudes and behavior survey) that when scored provide a single number will be used to determine the moderating effect of self efficacy, restraint and disinhibition maintaining diet and exercise changes
Change in humoral biomarkers of eating behavior | Weeks 0, 2, 4, 6, 8, 10, 12, 24
  The effect of diet and exercise on ghrelin, leptin, thyroid hormones, gut peptides, fatty acids
Gene expression profiles of glucose oxidation | Weeks 0, 2, 4, 6, 8, 10, 12, 24
  The effect of diet and exercise on gene expression profiles associated with glucose oxidation (i.e., hexokinase, phosphofructokinase, pyruvate dehydrogenase kinase 4, peroxisome proliferator-activated receptor alpha gene expression)
Gene expression profiles of fat oxidation | Weeks 0, 2, 4, 6, 8, 10, 12, 24
  The effect of diet and exercise on on gene expression profiles associated with fat oxidation (i.e., fatty acid translocase, fatty acid synthase, acetyl Co-A carboxylase 2, stearoyl Co-A desaturase gene expression)

OTHER OUTCOMES:
Single nucleotide polymorphisms (SNP) | Weeks 0
  Correlation of SNPs associated with skeletal muscle, catecholamine, executive function and food and exercise reinforcement
micro RNA (miRNA) | Weeks 0, 12, 24
  Correlation of miRNAs associated with skeletal muscle, executive function and food and exercise reinforcement

CONTACTS AND LOCATIONS:
Overall Officials: Shanon Casperson, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center; James Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT04577547/ICF_000.pdf